CLINICAL TRIAL: NCT03505528
Title: A Phase Ib Safety and Pharmacokinetics (PK)/ Pharmacodynamics (PD) Study to Determine the Dosage of Abraxane in Combination With Phenelzine Sulfate in Metastatic or Inoperable Locally Advanced Breast Cancer
Brief Title: An Early Phase Study of Abraxane Combined With Phenelzine Sulfate in Patients With Metastatic or Advanced Breast Cancer
Acronym: Epi-PRIMED
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EpiAxis Therapeutics (Industry)
Collaborators: The Canberra Hospital (Other); Southern Medical Day Care Centre (Unknown); Liverpool Cancer Therapy Centre (Other Government)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EpiAxis 001-0716
Record Dates: First submitted 2018-03-04; First posted 2018-04-23 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-07

CONDITIONS: Metastatic Breast Cancer
Keywords: Nanoparticle albumin-bound paclitaxel (Abraxane); Phenelzine Sulfate; Cancer stem cells; epigenetics; LSD1
MeSH Terms: conditions — Breast Neoplasms | interventions — Taxes; Albumin-Bound Paclitaxel; Phenelzine

STUDY DESIGN:
Intervention Model Description: An open, non-randomised, cumulative cohort group design (across 5 groups) with a target toxicity fraction of 30% and a margin of 10%. This means that a dose will be escalated between groups when the observed toxicity rate is < 20%, de-escalated when > 40% and maintained otherwise.
  The toxicity fraction is the number of participants receiving that dose who experience a DLT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cohort Group (Experimental): There are five patient cohort groups. Each will receive a progressively higher starting dose of phenelzine sulfate, consecutively. Cohort A will start at 15mg/day and will be increased to 30mg/d by week 2 and further increased to 45mg/d for week 3, which will be maintained throughout the study. Cohort B will start at 45mg/d and will be held constant throughout the Study. Similarly, Cohort C, D & E will start at 60, 75 and 90mg/d, respectively, and will also be held on this dose throughout the study. The decision to escalate the dose for the next cohort will be made on the basis of the number of dose limiting toxicity (DLT) events observed during the first 8 weeks in the preceding cohort group. In addition, all cohort groups will receive a constant dose of Abraxane at 100mg/m2.
  Interventions: Drug: Nanoparticle albumin-bound paclitaxel; Drug: Phenelzine Sulfate

INTERVENTIONS:
Drug: Nanoparticle albumin-bound paclitaxel — Abraxane is administered intravenous at a constant dose of 100mg/m2
  Other Names: Abraxane
Drug: Phenelzine Sulfate — Nardil is administered orally from a starting dose of 15mg/d to a maximum of 90mg/d
  Other Names: Nardil

SUMMARY:
This phase 1b study will determine the safety and efficacy of combined treatment of Abraxane and phenelzine sulfate (Nardil) for metastatic or locally advanced breast cancer.

Participants may be eligible to join this study if they are aged 18 years or above and have been diagnosed with metastatic breast cancer or inoperable locally advanced breast cancer.

All participants will receive a combination of intravenous Abraxane and an oral dose of phenelzine sulfate. Abraxane will be administered weekly for the first 3 weeks of a 4-week cycle for 3 consecutive cycles. Phenelzine sulfate will be taken daily for the duration of the 3 cycles. Five patient cohort groups will receive a progressively increasing dose of phenelzine sulfate. Safety and efficacy will be assessed weekly over the 3 cycles of treatment.

Although both drugs have been used in clinical care for more than a decade, they have not been intentionally combined together in a cancer therapy setting. This means that the combined effect of these two drugs has not been documented. This is being addressed in this study.

DETAILED DESCRIPTION:
Nanoparticle albumin-bound paclitaxel (Abraxane) will be administered intravenously over 3 cycles at a fixed dosage of 100mg/m2 to each study participant. This dose will be administered weekly for the first 3 consecutive weeks, over the 4 week cycle, before commencing the second and third cycles.

In addition to the fixed dose of nanoparticle albumin-bound paclitaxel, all patients will receive a continuous daily oral dose of phenelzine sulfate across all three cycles,

Each of the five patient cohort groups will receive a progressively higher starting dose of phenelzine sulfate, consecutively. Cohort A will start at 15mg/day and will be increased to 30mg/d by week 2 and further increased to 45mg/d for week 3, which will be maintained throughout the study. Cohort B will start at 45mg/d and will be held constant throughout the Study. Similarly, Cohort C, D & E will start at 60, 75 and 90mg/d, respectively, and will also be held on this dose throughout the study. The decision to escalate the dose for the next cohort will be made on the basis of the number of dose limiting toxicity (DLT) events observed during the first 8 weeks in the preceding cohort group.

Phenelzine sulfate compliance will be monitored weekly based on drug tablet returns.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are 18 years or older;
2. Fluent in written and spoken English and in a position to provide written informed consent to participate;
3. A patient who is in a position to attend a 12-week treatment regimen and end of study visit;
4. Metastatic Breast Cancer (MBC) or inoperable locally advanced breast cancer diagnosis based on pre-existing documented histopathology and medical imaging results, either Triple Negative Metastatic Breast Cancer (TNBC) or not;
5. Women with metastatic breast cancer or inoperable locally advanced breast cancer who have not received any cytotoxic therapy in the last 3 weeks;
6. Volunteers of child-bearing potential must have a negative serum pregnancy test (serum beta-human chorionic gonadotropin or ß-hCG) and have agreed to practice an effective, reliable contraceptive regimen for the duration of this clinical trial, such as an intrauterine device (IUD) or intrauterine system (IUS) with a failure rate of <1% stated on the product label or a male partner who is has been sterilised (vasectomy with documented azoospermia);
7. ECOG Performance Status 0 or 1; and
8. Adequate liver function as evidenced by bilirubin of <1.5 times upper limit of normal (ULN) and ALT/AST <2 times of ULN. However, AST and ALT of <5 times ULN if liver metastases are present.

Exclusion Criteria:

1. A patient who has been diagnosed as having HER2-positive metastatic breast cancer;
2. A concurrent condition that may limit the decision-making capabilities of the participant during the informed consent process;
3. A previous positive diagnosis of Human Immunodeficiency Virus (HIV) and/or Hepatitis C Virus (HCV) and/or Hepatitis B Virus (HBV) infection;
4. Women who are pregnant or lactating;
5. Uncontrolled, untreated intra-cranial metastases. However, controlled intra-cranial metastases are allowed, i.e. stable patients with more than a month after the completion of whole brain radiotherapy and not currently on steroids or anticonvulsants;
6. Current use of monoamine oxidase inhibitors (MOAI) or use of dextromethorphan
7. Current use of CNS depressants such as selective serotonin re-uptake inhibitors as well as specific medication for pain management including pethidine, tramadol, dextromethorphan, fentanyl and/or methadone. This includes the concurrent use of any serotoninergic agents or buspirone hydrochloride during the week preceding phenelzine sulfate administration, the active study treatment phase and the washout period at the end of study. Serotoninergic drugs may include but are not limited to the following: dexfenfluramine, fluoxetine, fluvoxamine, paroxetine, sertraline, citalopram and venlafaxine;
8. Previous use of nanoparticle albumin-bound paclitaxel;
9. Known allergy to phenelzine sulfate or similar MOAI; and
10. Known or suspected history of alcohol abuse;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) events | Assessed throughout the first 56 days
  The number of DLT events for nanoparticle albumin-bound paclitaxel and phenelzine sulfate combined, with the following events assessed using the NCI's CTCAE v4.3 toxicity criteria:
  * Grade 3 Febrile neutropenia;
  * Grade ≥2 peripheral neuropathy;
  * Any Grade 3 non-haematological toxicity except alopecia; nausea, vomiting, or diarrhoea for 72 hrs due to inadequate use of prophylaxis;
  * Grade 3 fatigue for > 7 days;
  * Non-hematologic Grade 3 or 4 laboratory AE that do not return to baseline or to Grade 1 within 7 days;
  * Grade 3 thrombocytopenia with signs of significant bleeding or platelet count Grade 4;
  * Blood bilirubin (total) Grade ≥3 for 72 hrs, AST or ALT Grade 3 for >7 consecutive days, AST or ALT Grade 4;
  * Persistent Grade 3 hypertension for >7 days & not responding to antihypertensive therapy or Grade 4 hypertension;
  * An inability to administer treatment (with >7 day delay) during Cycle 1 and Cycle 2 for toxicity reason; &
  * Any other treatment emergent SAE.

SECONDARY OUTCOMES:
Abraxane Cmax | Cmax will be assessed on two separate occasions. The first is at day 1 and is for the effect of nanoparticle albumin-bound paclitaxel alone. The second is at day 57 and is for the combined effect with phenelzine sulfate.
  To assess maximum plasma concentration (ng/ml) of nanoparticle albumin-bound paclitaxel alone and when combined with phenelzine sulfate.
Abraxane Tmax | Tmax will be assessed on two separate occasions. The first is at day 1 and is for the effect of nanoparticle albumin-bound paclitaxel alone. The second is at day 57 and is for the combined effect with phenelzine sulfate.
  To assess the time after infusion of nanoparticle albumin-bound paclitaxel alone and when combined with phenelzine sulfate to achieve peak maximum plasma concentration (minutes).
Abraxane Half-life | Half-life will be assessed on two separate occasions. The first is at day 1 and is for the effect of nanoparticle albumin-bound paclitaxel alone. The second is at day 57 and is for the combined effect with phenelzine sulfate.
  To assess the terminal half-life (minutes) of nanoparticle albumin-bound paclitaxel alone and when combined with phenelzine sulfate.
Abraxane AUC | AUC will be assessed on two separate occasions. The first is at day 1 and is for the effect of nanoparticle albumin-bound paclitaxel alone. The second is at day 57 and is for the combined effect with phenelzine sulfate.
  To assess the area under nanoparticle albumin-bound paclitaxel concentration time curve from 0 to infinity (ng minutes / ml) and when combined with phenelzine sulfate.
Nardil Cmax | Cmax will be assessed on day 57.
  To assess maximum plasma concentration (ng/ml) of phenelzine sulfate when combined with nanoparticle albumin-bound paclitaxel.
Nardil Tmax | Tmax will be assessed on day 57.
  To assess the time after ingestion of phenelzine sulfate, when combined with nanoparticle albumin-bound paclitaxel, to achieve peak maximum plasma concentration (minutes).
Nardil Half-life | Half-life will be assessed on day 57.
  To assess the terminal half-life (minutes) after ingestion of phenelzine sulfate, when combined with nanoparticle albumin-bound paclitaxel.
Nardil AUC | AUC will be assessed on day 57.
  To assess the area under Phenelzine Sulfate concentration time curve from 0 to infinity (ng minutes / ml) when combined with nanoparticle albumin-bound paclitaxel.
Circulating Tumour Cell (CTC) burden | CTC burden will assessed be at baseline and again at day 29, 57 and 85, whereas the CSC burden will assessed only at baseline and again at day 85.
  The CTC burden is expressed as the number of tumour cells observed per 30ml of blood.
PDL1 expressing Circulating Tumour Cell (CTC) burden | The PDL1 CTC expression burden will be assessed at baseline and again at day 29, 57 and 85, whereas the CSC burden will assessed only at baseline and again at day 85.
  The PDL1 expressing CTC burden is expressed as the number of CTC observed per 30ml of blood with PDL1 expression.
HER2 expressing Circulating Tumour Cell (CTC) burden | The HER2 CTC expression burden will be assessed at baseline and again at day 29, 57 and 85, whereas the CSC burden will assessed only at baseline and again at day 85.
  The HER2 expressing CTC burden is expressed as the number of CTC observed per 30ml of blood with PDL1 expression.
FFPE Tumour cells burden | Then burden will be assessed at baseline and again at day 85.
  The number of tumour cells observed per FFPE slide.
FFPE Stoma cells burden | Then burden will be assessed at baseline and again at day 85.
  The number of stoma cells observed per FFPE slide.
FFPE Cancer Stem Cells (CSC) burden | Then burden will be assessed at baseline and again at day 85.
  The number of CSC observed per FFPE slide.

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Yip, MBBS, Principal Investigator — ACT Health; Laeeq Malik, MBBS, Principal Investigator — ACT Health
Locations (3):
- Australia (3):
  - Canberra Region Cancer Centre, Canberra, Australian Capital Territory
  - Liverpool Cancer Therapy Centre, Sydney, New South Wales
  - Southern Medical Day Care Centre, Wollongong, New South Wales

IPD SHARING:
Plan to Share IPD: No
It is the sponsors intention to publish the aggregated study results after the completion of the study.

REFERENCES:
- [Background] Boulding T, McCuaig RD, Tan A, Hardy K, Wu F, Dunn J, Kalimutho M, Sutton CR, Forwood JK, Bert AG, Goodall GJ, Malik L, Yip D, Dahlstrom JE, Zafar A, Khanna KK, Rao S. LSD1 activation promotes inducible EMT programs and modulates the tumour microenvironment in breast cancer. Sci Rep. 2018 Jan 8;8(1):73. doi: 10.1038/s41598-017-17913-x. PMID 29311580
- [Background] Tan AHY, Tu W, McCuaig R, Hardy K, Donovan T, Tsimbalyuk S, Forwood JK, Rao S. Lysine-Specific Histone Demethylase 1A Regulates Macrophage Polarization and Checkpoint Molecules in the Tumor Microenvironment of Triple-Negative Breast Cancer. Front Immunol. 2019 Jun 12;10:1351. doi: 10.3389/fimmu.2019.01351. eCollection 2019. PMID 31249575
- [Derived] Prasanna T, Malik L, McCuaig RD, Tu WJ, Wu F, Lim PS, Tan AHY, Dahlstrom JE, Clingan P, Moylan E, Chrisp J, Fuller D, Rao S, Yip D. A Phase 1 Proof of Concept Study Evaluating the Addition of an LSD1 Inhibitor to Nab-Paclitaxel in Advanced or Metastatic Breast Cancer (EPI-PRIMED). Front Oncol. 2022 Jun 3;12:862427. doi: 10.3389/fonc.2022.862427. eCollection 2022. PMID 35719960
- See also: Sponsor's website — https://www.epiaxistherapeutics.com